CLINICAL TRIAL: NCT00413543
Title: Early Pulmonary Rehabilitation After Hospitalisation for Acute Exacerbation COPD
Brief Title: Pulmonary Rehabilitation for Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment insufficient: lack of motivated patients
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Jan W.K. van den Berg, pulmonologist, Isala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL11494.075.06
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; exacerbation; pulmonary rehabilitation; exercise tolerance; exacerbations; quality of life; readmissions
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interventional, rehabilitation (Experimental): 'early pulmonary lung rehabilitation'
  Interventions: Other: early pulmonary lung rehabilitation
- control (No Intervention): "standard care"

INTERVENTIONS:
Other: early pulmonary lung rehabilitation — early pulmonary rehabilitation, 10 days after discharge
  Arms: interventional, rehabilitation

SUMMARY:
This is a study to evaluate the effects of early pulmonary rehabilitation within 10 days after discharge from the hospital after a COPD exacerbation on exercise tolerance, exacerbations, re-admissions and the quality of life during 6 months.

DETAILED DESCRIPTION:
Study Design:

One hundred patients with an acute exacerbation of COPD admitted to the regular pulmonology department via the emergency room will be recruited after they have given written informed consent. Inclusion criteria are an age > 40 years or ≤ 80 years, at least 10 pack years of smoking history and COPD at least GOLD II. Each form of physical therapy is accepted outside pulmonary rehabilitation. Exclusion criteria include participation in a pulmonary rehabilitation program in the preceding year, comorbidity that can limit exercise training (for example: invalidating ischaemic heart disease, RA, malignancy and lung embolus), intolerance to prednisone, history of asthma, non-compliance, findings on chest radiography other than fitting with signs of COPD and a prior randomisation. During admission patients will receive standard exacerbation COPD treatment consisting of O2, combivent inhalation, antibiotics and prednisone. Exercise capacity is measured by a 6 minute walk test performed at discharge. The COPD GOLD classification is detected with a spirometry after completion of exacerbation therapy and before randomisation and discharge.

Both measurements are repeated after completion of the pulmonary rehabilitation program at 3 months. Quality of life is evaluated by the following questionnaires at discharge: St. George respiratory questionnaire (SGRQ), SF-36-scores (short form health survey) and clinical COPD questionnaire (CCQ). Before discharge, patients are randomised with a computer minimisation program for pulmonary rehabilitation or usual care with special attendance to age (< 70 years or ≥ 70 years), sex, length of hospital stay (< 7 days or ≥ 7 days), six minute walk test distance at discharge (< 100 or ≥ 100 meters) and predicted forced expiratory volume in one second (FEV1< or ≥ FEV1). Pulmonary rehabilitation will take place within ten days after discharge and shall be given by a multidisciplinary team (pulmonologist, respiratory nurse, physical therapist, dietician and a social worker). The program will last 2 hours weekly; 1 hour exercise training and one hour education during 8 weeks. All patients are followed up after discharge at 3 and 6 months. These questionnaires will be repeated after accomplishment of the pulmonary rehabilitation program at day 90 and day 180. Readmission rate will be also evaluated in this period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 40 years and < 80 years admitted to the hospital via ER
2. COPD at least Gold II
3. At least 10 pack years of smoking history
4. Physical therapy is tolerated, outside pulmonary rehabilitation

Exclusion Criteria:

1. Rehabilitation program < 1 year
2. Intolerance to prednisone
3. Non-compliance
4. Comorbidity limiting pulmonary rehabilitation
5. History of asthma
6. Prior randomisation
7. Findings on X thorax other than fitting with COPD

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance in meters | 2 years

SECONDARY OUTCOMES:
Exacerbations, readmissions and quality of life during follow-up | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Van den Berg, Dr., Study Director — Isala
Locations (1):
- Isala Klinieken, Zwolle, Overijssel, Netherlands